CLINICAL TRIAL: NCT03863665
Title: Prevention of Hypertensive Injury to the Brain by Intensive Treatment of Blood Pressure After Intracerebral Haemorrhage
Brief Title: Prevention of Hypertensive Injury to the Brain by Intensive Treatment of Blood Pressure After Intracerebral Haemorrhage (PROHIBIT-ICH)
Acronym: PROHIBIT-ICH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Imposed by the sponsor due to funding constraints
Sponsor: University College, London (Other)
Collaborators: University of Oxford (Other); The Stroke Association, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROHIBIT-ICH01
Record Dates: First submitted 2018-07-11; First posted 2019-03-05 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Intracerebral Hemorrhage
Keywords: Blood pressure; Hypertension; Secondary prevention
MeSH Terms: conditions — Cerebral Hemorrhage; Hypertension

STUDY DESIGN:
Intervention Model Description: Patients will be randomised in a 1:1 ratio to intervention or control arms of the study. Participants and their physicians will not be blinded to study arm allocation
Who Masked: Investigator, Outcomes Assessor
Masking Description: Researchers undertaking the neuroimaging analysis are masked to the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemetric Bluetooth-enabled home BP monitors (Experimental): Telemetric Bluetooth home BP monitors will be provided to participants during their inpatient stay or clinic visit, and will commence 3- times-daily readings immediately. The BP monitoring team will assess BP readings daily and advise medication adjustments to achieve a target BP of <120/80 mm Hg
  Interventions: Device: A&D BP Digital Blood Pressure Monitor (UA-767PBT-Ci) CE Declaration UA-767PBT-Ci
- Standard clinical care (No Intervention): Standard clinical care including usual BP treatment, without home monitoring, undertaken in the clinical care setting (primary and/or secondary care)

INTERVENTIONS:
Device: A&D BP Digital Blood Pressure Monitor (UA-767PBT-Ci) CE Declaration UA-767PBT-Ci — Telemetric home monitoring is a promising strategy to facilitate home BP monitoring after stroke, which should improve adherence and optimize medication to better control BP. Telemetry allows patients with hypertension to monitor their own BP and automatically send the information to a secure website, available to their clinicians to monitor and adjust their treatment.
  Arms: Telemetric Bluetooth-enabled home BP monitors

SUMMARY:
PROHIBIT-ICH will randomise participants (target=112) to compare a strategy of intensive blood pressure (BP) treatment (target <120/80 mm Hg) guided by remote telemetric home BP monitoring, versus standard primary care, in adult survivors of small vessel disease-related ICH. The investigators will establish the feasibility and safety of the intervention, the efficacy of BP reduction, and explore whether it reduces the progression of SVD-related injury on brain MRI.

DETAILED DESCRIPTION:
Eligible participants will be identified from acute stroke or high dependency units or outpatient clinics (neurology, geriatric, and neurosurgery) by a member of the research practitioner or member of research/clinical teams. Patients may be under the care of stroke physicians, geriatricians, neurologists, or neurosurgeons.

Baseline:

At baseline, the following trial specific procedures will be carried out after consent as a requirement for the study to commence:

* Medical history and demographic data recorded
* Blood pressure medication and dose recorded
* Blood pressure (BP), three seated office measures
* Blood test (venepuncture)
* MRI brain
* Cognitive assessment (Montreal Cognitive Assessment)
* Completion of an EQ-5D questionnaire
* 24-hour ABPM

Randomisation will be done using a web-based system in a 1:1 group assignment ratio to intensive remote telemetric home BP monitoring (RT-HBPM)-guided BP lowering (intervention group) or local primary care alone (control group), with stratification by ICH location (lobar versus non-lobar). In the intervention group, BP medication will adjusted on the basis of daily review of BP measures by the study physician in the central BP-monitoring team to target during 1-3 months to target a daily mean HBPM BP <120/80 mmHg.

Intervention:

The Telemetric Bluetooth home Blood Pressure-monitoring device will monitor participant's BP to keep the target of 120/80mm Hg, if this is not achievable then the BP medication will be adjusted accordingly in order to achieve a target of 120/80mm Hg at 3 months follow-up. BP readings (3 readings over 10-minutes in the seated position in the non dominant arm, unless hemiparesis) will be taken 3 times daily (early morning, early afternoon and evening). All BP data will be automatically transmitted centrally in real time to the device co-ordination site in Oxford. A dedicated research member will be responsible for checking all BP data daily on patients in the study, and will advise on adjusting medication according to a standard protocol based on the latest BHS guideline, to ensure that BP is lowered to the intervention arm target. The local study centre will send new prescriptions directly to patients (with communication simultaneously with the GP). For dose changes, advice will be given to participants by phone by the central study team. All medication changes will be notified to the local research team and GP; responsibility for BP treatment will be by the local PI.

Follow up:

3 month follow-up : completion of 3 month clinical data, blood pressure recorded and completion of Modified Cognitive assessment, EQ-5D questionnaire and home blood pressure acceptability questionnaire. 24-hour ABPM to be performed at the time of the 3 month follow-up visit.

12 month follow-up (Final visit): completion of 12 month CRF, blood pressure recorded, and completion of cognitive assessment and EQ-5D questionnaire. 24-hour ABPM to be performed at the time of the 12 month follow-up visit.

An MRI scan will be performed at baseline and the 12 month follow-up visit on all participants to identify markers of cerebral small vessel disease including:

* change in white matter hyperintensity volume
* change in white matter microstructure (DTI)
* change in the number of CMBs
* change in cerebral atrophy

Primary outcomes:

(a) BP study

(i) Acceptability: (a) ≥50% of eligible participants who were approached to participate agreed to be recruited; (b) <30% dropout from the intervention group (discontinuation of HBPM against the advice of the BP monitoring centre) prior to one month; (c) patient approval of the monitoring process in ≥70% of those who returned questionnaires.

(ii) Safety: between-group difference in number of serious adverse events related to reducing BP.

(iii) Efficacy: mean group difference in the change from baseline to 3-month follow-up assessment of systolic BP (mean of two sitting readings) in the intervention group versus the control group

(b) Imaging study

(i) Safety: evolution of new infarcts or ICH on 12-month follow-up MRI

(i) Efficacy: the progression on MRI white matter hyperintensity (WMH) volume (T2-weighted fluid-attenuated inversion recovery (FLAIR), or T2-weighted images when FLAIR was unavailable) between baseline and 12-month follow-up.

Secondary outcomes:

1. BP study: (i) between-group difference in mean daytime systolic BP change from baseline ABPM to 3-month ABPM; (ii) between-group differences at 3-month follow-up in assessment systolic BP and in mean daytime systolic BP on ABPM; (iii) between-group difference in number of BP-lowering drugs at follow-up; (iv) the maintenance of differences in BP after completion of centralised monitoring, assessed at 12-24-months follow-up.
2. Imaging study: neuroimaging outcomes including (but not limited to) the proportion of patients who develop new cerebral microbleeds (CMBs) over 1 year; number of new CMBs at 1 year; new infarcts or intracerebral haemorrhages at 1 year; change in mean diffusivity (MD), fractional anisotropy (FA) and other 3T DTI metrics; change in cerebral blood flow (CBF) on 3T PCASL; change in total brain volume, white matter volume and grey matter volume on 3T T1 volumetric images; composite neuroimaging measures (e.g summary SVD scores)

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥30 years) with spontaneous primary ICH (i.e. without known underlying structural, macrovascular or other cause (e.g. arteriovenous malformation, tumour) after adequate investigation at the discretion of the local investigator). This will include participants presumed to have cerebral SVD (both hypertensive arteriopathy and cerebral amyloid angiopathy)
2. Clinical team opinion that BP control since the ICH is not adequate AND the measured SBP prior to randomisation is ≥130 mm Hg
3. There is no time limit for recruitment; however, recruitment as soon as is practical after the ICH is encouraged. Recruitment at a later stage is acceptable as long as there is evidence of inadequate BP control AND SBP at randomisation is ≥130 mm Hg
4. Ability and willingness to undertake BP measurements,, either unassisted or with the help of a relative, friend or carer: this can be undertaken in any destination after hospital discharge (e.g. home, rehabilitation unit, nursing or care home)
5. Ability and willingness to attend and complete the study assessments including cognitive screen
6. Ability and willingness to provide informed consent, or with a suitable consultee available and able to participate in the intervention (e.g. with a motivated carer)

Exclusion Criteria:

1. Inability to provide informed consent or lack of suitable consultee (if unable to provide personal consent, lack of suitable consultee)
2. Evidence of a macrovascular or structural cause for ICH (e.g. AVM or tumour)
3. Diagnosis of dementia (DSM IV criteria, or self-reported or documented in medical records)
4. Low Functional status (MRS ≥4) before or after ICH or frailty likely to make participation in 1-year follow-up difficult for the participant
5. Life expectancy <2 years
6. Taking more than 2 BP-lowering medications (i.e. 3 or more) at the time of consent
7. Consistently good BP control (below 130/80 mm Hg on measures taken as part of routine clinical care) prior to planned recruitment, judged not to require more intensive treatment
8. Known flow-restricting intracranial/extracranial large arterial stenosis
9. Known absence of mobile phone coverage from all network operators and home internet at the participant's home
10. Known sensitivity or contra-indication to BP treatments (e.g. symptomatic postural hypotension) is not an absolute exclusion criterion, but more information must be provided
11. Note that participation in other CTIMP or device trial is NOT an automatic exclusion criterion

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2023-04-29 (Actual)

PRIMARY OUTCOMES:
BP Study: Efficacy | 3 months from randomisation
  Magnitude of difference in assessment BP at 3 months in the intervention arm versus the control arm compared with baseline measures
BP Study: Feasibility | 3 months from randomisation
  At least ≥50% of eligible participants agree to participate, <30% dropout from the intervention arm (discontinuation of home BP monitoring against the advice of the BP monitoring centre) prior to 1 month, Patient approval of the monitoring process in ≥70% of those randomised to the intervention arm.
BP Study: Safety | 3 months from randomisation
  Serious adverse events related to reducing BP in intervention arm
Imaging Study: Efficacy | 12 months from randomisation
  Progression in MRI white matter hyperintensity (WMH) volume since baseline
Imaging Study: Safety | 12 months from randomisation
  Evolution of new infarcts or ICH on 12-month follow-up MRI

SECONDARY OUTCOMES:
Incidence of recurrent vascular events | 12 months from randomisation
  Any incidence of vascular events reported in both arms
Cognitive ability assessed by the Cognitive Assessment (MoCA) questionnaire in both arms | 12 months from randomisation
  The Cognitive Assessment is a questionnaire widely used as a screening assessment for detecting cognitive impairment. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. An abbreviated version of the assessment assessing attention, verbal learning, memory, executive functions/language and orientation can be performed over the phone.
The number of BP lowering drugs at 3 months and at 1 year follow-up visits | 12 months from randomisation
  This will detected in both arms and compared
Mean daytime BP at 1 year on 24-hour ABPM | 12 months from randomisation
  The blood pressure measured in both groups
Neuroimaging outcomes: the proportion of patients who develop new cerebral microbleeds (CMBs) over 1 year | 12 months from randomisation
  neuroimaging outcomes will be measured in both arms
Neuroimaging outcomes: the proportion of patients who develop new infarcts or intracerebral haemorrhages at 1 year | 12 months from randomisation
  neuroimaging outcomes will be measured in both arms
Neuroimaging outcomes: measure change in mean diffusivity (MD) | 12 months from randomisation
  neuroimaging outcomes will be measured in both arms
Neuroimaging outcomes: measure fractional anisotropy (FA) | 12 months from randomisation
  neuroimaging outcomes including (but not limited to) ; ; change in mean diffusivity (MD), fractional anisotropy (FA) and other 3T DTI metrics; change in cerebral blood flow (CBF) on 3T PCASL; change in total brain volume, white matter volume and grey matter volume on 3T T1 volumetric images; composite neuroimaging measures (e.g summary SVD scores)
Neuroimaging outcomes: measure change in brain volume | 12 months from randomisation
  neuroimaging outcomes including (but not limited to) : change in cerebral blood flow (CBF) on 3T PCASL; change in total brain volume, white matter volume and grey matter volume on 3T T1 volumetric images; composite neuroimaging measures (e.g summary SVD scores)

CONTACTS AND LOCATIONS:
Overall Officials: David Werring, Study Chair — University College, London
Locations (16):
- United Kingdom (16):
  - Royal United Hospitals Bath, Bath
  - West Suffolk Hospital, Bury St Edmunds
  - Cambridge, Cambridge
  - Edinburgh, Edinburgh
  - Glasgow, Glasgow
  - King's, London
  - St George's, London
  - Imperial, London
  - UCLH, London
  - Croydon University Hospital, London
  - Luton & Dunstable Hospital, Luton
  - Nottingham, Nottingham
  - Oxford, Oxford
  - Royal Preston, Preston
  - Salford, Salford
  - Sheffield, Sheffield

REFERENCES:
- [Derived] Li L, Poon MTC, Samarasekera NE, Perry LA, Moullaali TJ, Rodrigues MA, Loan JJM, Stephen J, Lerpiniere C, Tuna MA, Gutnikov SA, Kuker W, Silver LE, Al-Shahi Salman R, Rothwell PM. Risks of recurrent stroke and all serious vascular events after spontaneous intracerebral haemorrhage: pooled analyses of two population-based studies. Lancet Neurol. 2021 Jun;20(6):437-447. doi: 10.1016/S1474-4422(21)00075-2. PMID 34022170

DOCUMENTS (1):
  • Study Protocol (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/65/NCT03863665/Prot_000.pdf